CLINICAL TRIAL: NCT02208817
Title: Development of a Novel Paediatric Continuous Early Warning Monitor for the Children at Risk of Respiratory and Cardiovascular Collapse - The Paediatric Refill Study (PRefill)
Brief Title: The Paediatric Refill Study (PRefill)
Acronym: PRefill
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 14021; MRK0076101 (Other Grant/Funding Number: Medical Research Council)
Record Dates: First submitted 2014-07-14; First posted 2014-08-05 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Septicaemia; Deformity of Spine; Trauma
Keywords: capillary refill; paediatric early warning score; photoplethysmography
MeSH Terms: conditions — Toxemia; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Ill patients: Ill patients who require Paediatric Intensive Care or Paediatric High Dependency Care
- Well Controls: Matched controls who are well (PEWS<3)
- Parent feedback: Feedback from parents/carers of children recruited into the PRefill study
- Healthcare professionals feedback: Feedback from healthcare professionals who have cared for a child with the device on

SUMMARY:
2 recent national reports 'Why Children Die' and 'Are we there yet?'identified deficiencies in recognising and managing sick children. Key recommendations from both reviews included the development and adoption of 'track and trigger' or a paediatric early warning score (PEWS) to better identify the sick or deteriorating child. PEWS tools offer the potential to identify and respond sooner to clinical deterioration. Capillary refill time (CRT) is a measure of skin blood flow and is a vital part of many early warning and resuscitation scores. It is a sensitive marker of infection and dehydration in children. However, due to how it is performed and interpreted CRT is prone to marked variability between observers.

We have Medical Research Council (MRC) funding to develop an automated capillary refill device and user interface to provide a paediatric continuous early warning (PaedCEW) monitoring system. The PaedCEW system would complement and support current clinical practice and aim to address the difficulties of recognising ill children.

We aim to recruit 20 ill children on the Paediatric Intensive Care Unit (PICU) with 2 matched controls without significant illness from the Nottingham Children's Hospital. The 20 ill children will have their CRT (and PaedCEW score) monitored before, during and after admission to PICU. This will allow correlation with invasive (BP, central venous oxygen saturations, lactate) and noninvasive (CRT, heart rate, cardiac output) measures of cardiovascular status during periods of stability and compromise. Matched controls will be monitored for around 24 hours. This pilot study will allow development of our system.

This is a proof of concept study. This study aims to demonstrate a novel device for measuring CRT. Its correlation with noninvasive measures of cardiovascular status will enable a pragmatic comparison with current clinical practice. In addition, correlation with invasive measures of cardiovascular status will enable us to calculate sensitivity, specificity, negative predictive value (NPV) and positive predictive value (PPV).

DETAILED DESCRIPTION:
Following recruitment, patients will have two devices placed on their skin, one on a limb (e.g. forearm), and one on their chest. They will be fixed to the skin using medical adhesive tape. The devices will be left on for around 1 hour on the "well patients" who are on a general paediatric ward. At the end of this time a member of the research team will remove the devices.

For patients going to the paediatric intensive care unit (PICU) the devices will be used to gather the CRT data before admission (where possible), during and following discharge from the PICU. The PICU participants will have the device left on during their stay, with the agreement of the clinical team caring for the patient, with the device being resited every 4-6 hours as is normal practice for medical devices attached to the skin. Data will be collected in this way during the PICU stay (which is typically 2-3 days) or until the patient is transferred to the general ward. Before they go home, these participants will be monitored again for up to an hour with the CRT devices to obtain data when they are well.

Collecting data in this way should allow us to show that our CRT device can detect a 30% difference in perfusion between the well and the unwell patient. By comparing well patient to unwell patient, and by comparing unwell patient, with themselves when well. For each participant we will collect routine demographic details, medical history details, Fitzpatrick skin colour assessment (that is their skin tone according to a recognised scale), height, weight and vital signs. Where taken, we will collect clinically relevant data in relation to the treatment received and results of clinical investigations for correlation with our device data. Patients on the PICU will have noninvasive measures of perfusion performed by the clinical team. The research team will also perform these at agreed times suitable to the care of the patient. This will include capillary refill and ultrasound assessment of blood flow (cardiac output).

We will also conduct a semistructured interview with the patient and/or their parents/carer at the time of the study to gain feedback on the device. This should take about 15 minutes and will take the form of a semistructured interview. We will also seek user (i.e. healthcare professionals) feedback on the device and the accompanying GUI using a semistructured interview (approximately 15 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Children & Young Adults
* Patients aged 1 month to 15 years with parental or legal guardian written informed consent.
* Patients groups:
* Patients who require PICU or high dependency care
* Matched controls who are well (PEWS<3)
* Must have a realistic prospect of survival
* Parents/carers (for the interview element of the study):
* Parents/carers of children recruited into the PRefill study
* Healthcare professionals (for the interview element of the study):
* Healthcare professionals who have cared for a child with the device on

Exclusion Criteria:

* Children & Young Adults
* Known pregnancy
* Underlying cardiac anomaly likely to affect perfusion,
* PEWS ≥3 (in matched well controls)
* Severe eczema/burns/other skin condition on site where CRT device needs to be positioned
* Known allergy to medical adhesive
* Parents/carers (for the interview element of the study):
* Unable to communicate despite translation services
* Healthcare professionals (for the interview element of the study)
* None

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children will be recruited in The Queens Medical Centre, Nottingham University Hospitals NHS Trust, a teaching hospital, which has a paediatric intensive care unit (PICU).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2014-08; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Detect a 30% difference in measured CRT value between well children (PEWS <3, with normal perfusion) and unwell children (PEWS ≥3, with reduced perfusion). | Exit from study; Well patients within 1-2 hours; Unwell patients after leaving PICU average 3 days

SECONDARY OUTCOMES:
i.Feedback on acceptability of the device from patients, carers/parents, and healthcare professionals, and feedback on the graphical user interface (GUI) from healthcare professionals. | on completion of feedback, 30 minutes
ii. Correlation of automated CRT results with vital cardiovascular clinical observations and tests - both invasive and non-invasive. | During study phase average 3 days
iii. Correlation of automated CRT results with treatments supporting the cardiovascular and neurological system | during study phase average 3 days
CRT in well compared with unwell patients | Grouped at end of study 12 months
CRT changes with age and ethnicity in well children | grouped at end of study 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Don Sharkey, PhD, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham Univeristy Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom